CLINICAL TRIAL: NCT05919524
Title: Fractionated Stereotactic Ablative Body Radiotherapy (SBRT) With FOcal Dose Escalation on Dominant Lesion in Localized Prostate Cancer
Brief Title: SBRT With Focal Dose Escalation on DIL in Localized Prostate Cancer
Acronym: SAFO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Almudena Zapatero (Other)
Responsible Party: Sponsor-Investigator, Almudena Zapatero, Principal Investigator and Sponsor, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT Focal SAFO
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT with mpMRI guided focal boost (Experimental): SBRT 36.25 Gy in 5 sessions of 7.25 Gy to the entire prostate (including seminal vesicles) with a DIL simultaneous integrated focal boost (SIB) up to 50 Gy in 5 sessions, with partial protection of the prostatic urethra and bladder trigone.
  Interventions: Radiation: Prostate SBRT (stereotactic body radiation therapy) with focal boost

INTERVENTIONS:
Radiation: Prostate SBRT (stereotactic body radiation therapy) with focal boost — * Prostate SBRT delivered to a dose of 36.25 Gy in 5 fractions of 7.25 Gy to the entire prostate (including seminal vesicles) using VMAT
  * mpMRI defined DIL was simultaneously boosted up to 50 Gy in 5 sessions to the mpMRI identified DIL.
  * Additional urethra and bladder trigone sparing constrains
  * Daily IGRT with cone beam CT and intrafraction gold-seeds fiducial tracking
  Other Names: SABR with SIB; SBRT focal intensification

SUMMARY:
Stereotactic ablative Body Radiotherapy (SBRT) is an advanced radiation technique that allows for precise delivery of higher radiation doses in fewer treatment sessions, resulting in a shorter overall treatment duration. The available clinical evidence suggests that SBRT is highly effective in controlling localized prostate cancer (PCa) with acceptable side effects.

On the other side, dose escalation is a commonly employed strategy in radiotherapy for prostate cancer. Recent studies have confirmed a dose-response relationship, demonstrating improved biochemical control with focal dose escalation to the identified dominant intraprostatic lesion (DIL) on multiparametric magnetic resonance imaging (mpMRI) of the prostate.

The hypothesis of this study is that the combination prostate SBRT with focal dose intensification on the DIL with preservation of the prostatic urethra, would lead to a higher probability of local control without a significant increase in toxicity compared to standard clinical practice.

This is a prospective single-arm phase II study designed to evaluate the effectiveness, safety and impact on quality of life of focal dose intensification using SBRT technology and extreme hypofractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Primary localized PCa, cN0 and cM0, intermediate or high-risk disease according to NCCN 2023
* Signed written informed consent for this study
* T2-T3a clinical stage with visible DIL on mpMRI
* ECOG 0-1
* Desirable prostate volume (not mandatory) < 80 cc or > 80 cc if urinary function is preserved and dosimetrically feasible
* IPSS ≤ 18 (International Prostate Symptom Score)

Exclusion Criteria:

* Unresolved previous prostatitis, symptomatic urethral stenosis
* Bilateral hip prosthesis
* T3b-4 clinical stage or N1
* M1 (presence of distant metastases)
* Previous surgery at the prostate level (Transurethral Resection of the Prostate) within the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical progression-free survival | 3 years
  Biochemical progression as Phoenix definition (PSA nadir +2 ng/ml)
Local control | 12 months
  Disappearance of suspicious image on mpMRI.

SECONDARY OUTCOMES:
Incidence and severity of acute urinary treatment-related adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale | 90 days
  Every urinary event occurring within 3 months from treatment completion will be defined as "acute event".
  All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Incidence and severity of acute rectal treatment-related adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale | 90 days
  Every rectal event occurring within 3 months from treatment completion will be defined as "acute event".
  All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Incidence and severity of late urinary treatment-related adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale | 2 years
  Every urinary event occurring after 3 months from treatment completion will be defined as "late event".
  All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Incidence and severity of late rectal treatment-related adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale | 2 years
  Every rectal event occurring after 3 months from treatment completion will be defined as "late event".
  All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Patient reported outcomes and quality of life assessment | 2 years
  Impact on Quality of life affecting the genitourinary, gastrointestinal, sexual and hormonal domains using the EPIC-26 short form (International Prostate Symptom Score (IPSS) and Expanded Prostate Index Composite-26

CONTACTS AND LOCATIONS:
Locations (1):
- La Princesa University Hospital, Health Research Institute, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Zapatero A, Castro P, Roch M, Carnero PR, Carroceda S, Rosciupchin AES, Hernandez SH, Cogorno L, Iturriaga AG, Garcia DB. Functional imaging guided stereotactic ablative body radiotherapy (SABR) with focal dose escalation and bladder trigone sparing for intermediate and high-risk prostate cancer: study protocol for phase II safo trial. Radiat Oncol. 2024 May 3;19(1):54. doi: 10.1186/s13014-024-02440-7. PMID 38702761